CLINICAL TRIAL: NCT00967928
Title: Phase I Everolimus Dose Finding Study for the Treatment of Stage IV or Recurrent, Non-resectable, Cervical Cancer With Standard Whole Pelvic Radiation Therapy in Combination With Weekly Cisplatin and Daily Everolimus
Brief Title: Everolimus Dose Finding Study for Stage IV or Recurrent Cervical Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATDTCC0801
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Cervical Cancer
Keywords: Stage IV or Recurrent Cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Everolimus; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental): All subjects receive RAD001 in combination with standard field whole pelvic radiation and cisplatin.
  Interventions: Drug: RAD001; Drug: Cisplatin; Radiation: External Beam Whole Pelvis Radiation Therapy

INTERVENTIONS:
Drug: RAD001 — RAD001 will be administered orally as 5 mg qod, 5 mg qd, or 10mg qd continuously from study Day 1 until the end of whole pelvic radiation therapy unless the patient develops progression of disease or unacceptable toxicity prior to that.
  Other Names: Afinitor; Everolimus
Drug: Cisplatin — Cisplatin will be administered intravenously once weekly at 40mg/m2 for 6 weeks. The preferred administration day is Monday.
  Other Names: CDDP; Platinol
Radiation: External Beam Whole Pelvis Radiation Therapy — Patients will receive 180 cGy daily fraction Monday through Friday x 25 days (4500 cGy total) using a four field technique throughout the entire treatment with all fields treated each day.

SUMMARY:
This Phase 1, single-site, dose-escalation study is being conducted to determine the maximum tolerated dose (MTD) of RAD001 as part of a specified combination regimen.

DETAILED DESCRIPTION:
This Phase 1, single-site, dose-escalation study is being conducted to determine the MTD of RAD001 as part of a specified combination regimen. The combination regimen will be standard field whole pelvic RT in combination with cisplatin at 40mg/m2 weekly with RAD001 at dose escalation daily starting at 5 mg qod, then 5 mg qd, then 10 mg qd during the period of whole pelvic radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have at least one measurable site of disease according to Response Evaluation Criteria in Solid Tumors criteria that has not been previously irradiated.
* Female patient aged ≥18 years.
* Patient has life expectancy of at least 12 weeks at study start.
* Patient has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at study start.
* Patient has diagnosis of stage IV or recurrent, non-resectable, cervical cancer at study start.
* Patient has received no prior chemotherapy.
* Patient has adequate hematologic function:

  * Absolute neutrophil count [ANC] ≥1500/μL
  * Platelets ≥100,000/μL
  * Hemoglobin > 9g/dL
* Patient has adequate renal function:

  * Serum creatinine ≤ 2.0 mg/dL
  * Calculated creatinine clearance ≥ 50 mL/min
* Patient has adequate hepatic function:

  * Serum bilirubin ≤1.5 x ULN
  * ALT and AST ≤2.5 × ULN (≤ 5 x ULN in patients with liver metastases)
* INR <1.5 (or < 3 on anticoagulants)
* Patient has fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN.
* Patient is able to provide signed informed consent.

Exclusion Criteria:

* Patient has neuroendocrine or small cell carcinoma of the cervix.
* Patient has previously used any biologic therapy with VEGF, VEGFR, or ErbB1/ErbB2 inhibitors.
* Patient is currently receiving anticancer therapies or has received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.).
* Patient has had a major surgery or significant traumatic injury within 4 weeks of start of study drug; patient has not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patient might require major surgery during the course of the study.
* Patient has had prior treatment with any investigational drug within the preceding 4 weeks before study start.
* Patient is receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period. Patients should also avoid close contact with people who have received live vaccines during treatment with everolimus. Examples of live vaccines are: intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, and TY21a typhoid vaccines.
* Patient has known brain or leptomeningeal metastases.
* Patient has had other malignancies within the past 3 years except for adequately treated squamous cell carcinomas of the skin.
* Patients has any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Symptomatic congestive heart failure of New York Heart Association Class III or IV.
  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.
  * Severely impaired lung function defined as spirometry and diffusing capacity (DLCO) that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air.
  * Uncontrolled diabetes as defined by fasting serum glucose >1.5 × ULN.
  * Active (acute or chronic) or uncontrolled severe infections.
  * Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
* Patient has a known history of human immunodeficiency virus seropositivity.
* Patient has impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
* Patient has an active, bleeding diathesis.
* Female patient who is pregnant or breast feeding, or an adult of reproductive potential who is not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial and for up to 8 weeks after ending treatment by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of RAD001.)
* Patient has received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* Patient has a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients.
* Patient has history of noncompliance to medical regimens.
* Patient is unwilling to or unable to comply with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose for RAD001 as adjunct therapy to standard upfront treatment of advanced stage cervical cancer in combination with weekly cisplatin and whole pelvic external beam radiation | every 7 days
To determine the dose limiting toxicities for RAD001 as adjunct therapy to standard upfront treatment of advanced stage cervical cancer in combination with weekly cisplatin and whole pelvic external beam radiation | every 7 days

SECONDARY OUTCOMES:
To determine the pharmacokinetics of RAD001 given as adjunct therapy to standard upfront treatment of advanced stage cervical cancer | day 1 and day 15 during study treatment
To evaluate the pharmacogenetics of RAD001 in the specified patient population | day 1 prior to starting study treatment
To evaluate microvessel density pre-and post-treatment with the specified treatment regimen in the specified patient population | day 1 and end of treatment
To evaluate potential correlations between biomarkers HIF-1a, TSP-1, P53, VEGF, and VEGFR and use of the specified treatment regimen in the specified patient population | day 1 and end of treatment
To evaluate progression free survival in the specified patient population | from the time of treatment start until progression or up to 5 years after completion of study treatment
To assess quality of life as indicated by the Patient Care Monitor in the specified patient population | every 7 days during study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Todd D Tillmanns, MD, Principal Investigator — The West Clinic